CLINICAL TRIAL: NCT00518947
Title: Pharmacotherapy of Treatment-Resistant Mania
Acronym: TRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01MH050634 (NIH)
Record Dates: First submitted 2007-08-08; First posted 2007-08-21 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Mania
Keywords: Bipolar Disorder; Mania; Antimanic; Verapamil; Lithium
MeSH Terms: conditions — Mania; Bipolar Disorder | interventions — Lithium; Verapamil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Continued-Lithium
  Interventions: Drug: Lithium
- 2. (Experimental): Verapamil
  Interventions: Drug: verapamil
- 3. (Experimental): Verapamil plus Lithium
  Interventions: Drug: verapamil plus lithium

INTERVENTIONS:
Drug: Lithium — Treatment with lithium carbonate was initiated at a dose of 900-1200 mg/day. Serum lithium levels were monitored twice weekly, and the dose was adjusted to attain target levels between 0.8 and 1.0 mmol/L by the end of week one, with subsequent levels as high as 1.4 mmol/L permitted if needed.
  Arms: 1
Drug: verapamil — The initial dose of verapamil was 80 mg b.i.d., and this was raised by 80 mg/day every three days to a maximum of 480 mg/day, unless intolerable side effects were produced at a lower level, in which case the dose was maintained at the highest tolerated amount.
  Arms: 2.
Drug: verapamil plus lithium
  Arms: 3.

SUMMARY:
Verapamil has been found in some but not all studies to have antimanic activity. Therefore, we investigated the use of verapamil, alone or as an adjunctive treatment, in manic patients who did not respond to an initial adequate trial of lithium. Each study phase lasted three weeks. Subjects were treated openly with lithium in Phase 1 (n=45). Those who failed to respond were randomly assigned to double-blind treatment in Phase 2 with either verapamil (n=10) or continued lithium (n=8). Phase 2 responders were continued on the same medication in Phase 3. Phase 2 nonresponders (n=10) were assigned to combined verapamil/lithium in Phase 3.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients were required to have a lifetime diagnosis of bipolar 1 or schizoaffective disorder, a current manic episode meeting DSM-IV criteria, and ratings >/= 7 on the Raskin Severity of Mania Scale and >/= 15 on the Bech-Rafaelsen Mania Scale.

Exclusion Criteria:

Patients were excluded if they had:

* A pattern of severe rapid-cycling in which the patient consistently failed to meet the duration criteria for discreet episodes of syndromal mania or depression according to DSM-IV
* Sustained drug or alcohol abuse within the past three years
* Schizophrenia
* Organic affective syndrome
* A presenting episode that was secondary to the effect of any pharmacologic agent
* The presence of significant medical illness that would preclude or unduly complicate the intended pharmacologic management of the episode
* In females, refusal to use appropriate contraception; or
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1994-11; Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
A > 50% reduction in Bech-Rafaelsen Mania Scale score (relative to the baseline score at the start of the phase), and, a total Bech-Rafaelsen Mania Scale score < 11 | 3 weeks
Very much improved or much improved (compared to baseline) on the Clinical Global Impressions scale | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan G. Mallinger, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Frank E, Kupfer DJ, Gerebtzoff A, Meya U, Laghrissi-Thode F, Grochocinski VJ, Houck PR, Mallinger AG, Gibbons RD. The development of study exit criteria for evaluating antimanic compounds. J Clin Psychiatry. 2001 Jun;62(6):421-5. doi: 10.4088/jcp.v62n0604. PMID 11465518
- [Result] Mallinger AG, Thase ME, Haskett R, Buttenfield J, Luckenbaugh DA, Frank E, Kupfer DJ, Manji HK. Verapamil augmentation of lithium treatment improves outcome in mania unresponsive to lithium alone: preliminary findings and a discussion of therapeutic mechanisms. Bipolar Disord. 2008 Dec;10(8):856-66. doi: 10.1111/j.1399-5618.2008.00636.x. PMID 19594501